CLINICAL TRIAL: NCT04123470
Title: A Phase I/II Trial Investigating LOAd703 in Combination With Atezolizumab in Malignant Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lokon Pharma AB (Industry)
Collaborators: Precision Oncology LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LOKON003; 2019-003300-12 (EudraCT Number)
Record Dates: First submitted 2019-10-09; First posted 2019-10-11 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — atezolizumab

STUDY DESIGN:
Intervention Model Description: Participants treated with LOAd703 at two dose levels (1x10e11 VP and 5x10e11VP) and fixed dose of atezolizumab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Delolimogene mupadenorepvec plus atezolizumab
  Interventions: Genetic: delolimogene mupadenorepvec; Biological: atezolizumab

INTERVENTIONS:
Genetic: delolimogene mupadenorepvec — LOAd703 is an oncolytic adenovirus encoding TMZ-CD40L and 4-1BBL
  Other Names: LOAd703
Biological: atezolizumab — Atezolizumab is an anti-PD-L1 antibody

SUMMARY:
This study aims to evaluate safety and effect of combining an oncolytic adenovirus (delolimogene mupadenorepvec; LOAd703) with atezolizumab in patients with melanoma. LOAd703 will be administered intratumorally for up to 12 injections while atezolizumab will be administered intravenously for the duration of the active study visits (up to 57 weeks). The patients are then monitored for survival for maximum study participation of 48 months. The treatments will be given every 3 weeks. The patients will then be monitored for toxicity, PK, ADA, immune responses, virus shedding, tumor response by RECIST 1.1 and survival.

DETAILED DESCRIPTION:
This is a single arm, open-label, multicenter trial. This study aims to evaluate safety and effect of combining an oncolytic adenovirus (delolimogene mupadenorepvec; LOAd703) with atezolizumab in patients with melanoma. Patients will receive up to 12 LOAd703 intratumoral treatments in combination with intravenous infusions of atezolizumab. LOAd703 will be tested at two dose levels to determine the maximum tolerated dose (MTD) of LOAd703 evaluated in the study using a BOIN design. The LOAd703 dose can be divided for intratumoral injection into as many as 3 tumor lesions. Atezolizumab will be tested at a fixed dose. At least 25 response evaluable patients will be enrolled at the MTD for evaluation of their response using binominal testing. The maximum number of evaluable patients in the study is 35. The patients will then be monitored for toxicity, PK, ADA, immune responses, virus shedding, tumor response by RECIST 1.1 and survival.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological confirmation of melanoma.
2. A life expectancy of at least 3 months as per the investigator
3. Valid for Swedish patients: Patients has locally advanced melanoma or metastatic melanoma, but not eligible for complete resection of melanoma Valid for US patients: Patients has locally advanced melanoma or metastatic melanoma.
4. The patient has measurable disease (e.g., measurable tumor lesions must be present that can accurately be measured in at least one dimension with a minimum size of 10 mm by CT scan and MRI, 10 mm caliper measurement by clinical exam (when superficial), and/or 20 mm by chest X-ray).
5. Patient has at least one injectable tumor lesion that has not been irradiated or has been irradiated but disease progression documented at the site subsequent to radiation therapy.
6. The patient has received appropriate treatment with an anti-PD-1 or anti-PD-L1 antibody with or without an anti-CTLA4.
7. Valid for Swedish patients: Patients whose advanced melanoma has a B-Raf mutation must have received appropriate therapy with tyrosine kinase inhibitor(s) and/or MEK inhibitor Valid for US patients: Patients whose advanced melanoma has a B-Raf mutation may have received appropriate therapy with tyrosine kinase inhibitor(s) and/or MEK inhibitor as assessed by the investigator.
8. Age ≥ 18 years.
9. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
10. Serum albumin ≥ 2.5 mg/dL.
11. Absolute neutrophil count (ANC) ≥1.0 x 10e9/L.
12. Platelet count ≥ 100 x 10e9/L.
13. Prothrombin (INR) ≤ 1.5 or prothrombin time (PT) ≤ 1.5 times ULN; and either partial thromboplastin time or activated partial thromboplastin time (PTT or aPTT) ≤ 1.5 times the ULN.
14. Bilirubin < 1.5 times the institutional upper limit of normal (ULN).
15. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 (≤ 5 if liver metastases are present) times the institutional ULN.
16. The patient must have signed informed consent.

Exclusion Criteria:

1. Malignant melanoma that is uveal.
2. Subjects considered by the investigator to have rapid clinical progression due to melanoma
3. Subjects must not have greater than 3 cerebral melanoma metastases, and/or clinically active cerebral melanoma metastases, and/or a requirement for corticosteroid therapy, and/or carcinomatous meningitis regardless of clinical stability.
4. Any concurrent treatment that would interfere with the effect mechanisms of atezolizumab and LOAd703, including, but not limited to, continuous high-dose corticosteroids (>10 mg per day), lymphodepleting antibodies, or cytotoxic agents.
5. Treatment with inhibitors of immune function, such as lymphotoxic monoclonal antibodies (e.g., alemtuzumab), or rapamycin/rapamycin analogs, or cytotoxic agents within 21 days of the first dose of LOAd703/atezolizumab.
6. Therapeutic treatment with systemic antibiotics within 14 days of the first dose of LOAd703/atezolizumab.
7. Treatment with biologic therapy within 21 days of the first dose of LOAd703/atezolizumab.
8. Treatment with cytotoxic anticancer therapy within 14 days of the first dose of LOAd703/atezolizumab.
9. Treatment with wide-field radiation within 14 days of the first dose of LOAd703/atezolizumab.
10. Prior treatment with an adenovirus-based gene therapy.
11. Use of any investigational agents within 21 days of the first dose of LOAd703/atezolizumab.
12. The use of systemic immunostimulatory agents (including, but not limited to, interferons and IL2) are prohibited within 21 days or 5 half-lives (whichever is longer) of the first dose of LOAd703/atezolizumab.
13. Failed resolution/improvement of AEs including those related to anti-PD-1/anti-PD-L1 to grade 0-1 and requirement for treatment with >10 mg/day prednisone (or equivalent) for at least two weeks prior to registration.
14. History of CTCAE grade 4 immune-related AEs from monotherapy using an anti-PD-1/anti-PD-L1 antibody.
15. History of CTCAE grade 4 AE that require steroid treatment (>10 mg/day prednisone or equivalent) for >12 weeks.
16. Patients requiring warfarin are not eligible (low molecular weight heparin is permitted).
17. Women who are pregnant (as confirmed by pregnancy test during screening in applicable patients), breastfeeding, or planning to become pregnant during the study period, or women of childbearing potential who are not using acceptable highly effective contraceptive methods. A woman is considered of childbearing potential if she is not surgically sterile or is less than 1 year since her last menstrual period. The following are acceptable as highly effective contraceptive methods: combined (estrogen- and progesterone-containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progesterone-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion and vasectomized partner or abstinence of heterosexual intercourse during the entire study period (depending on the preferred and usual life style of the subject).
18. Men who do not consent to the use of condoms during intercourse during study participation or has a partner of childbearing potential, who will not use any of the highly effective contraceptive methods exemplified in exclusion criteria no 18.
19. Known active hepatitis B or C infection, or HIV infection.
20. Patients with active, severe autoimmune disease or immune deficiency or previous Guillain-Barré syndrome. Patients with eczema, psoriasis, lichen simplex chronicus or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

    1. Rash must cover <10% of body surface area.
    2. Disease is well-controlled at baseline and requires only low-potency topical corticosteroids.
    3. Occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months.
21. History of leptomeningeal disease.
22. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently).
23. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan or tested reduced functional respiration capacity. However, history of radiation pneumonitis in the radiation field (fibrosis) is permitted.
24. Unstable angina, uncontrolled cardiac arrhythmia, recent (within 3 months) history of myocardial infarction or stroke, or New York Class III/IV congestive heart failure.
25. Major surgical procedure other than for the malignant melanoma diagnosis, within 4 weeks prior to initiation of the study treatment, or anticipation of the need for a major surgical procedure during the study.
26. Prior allogeneic stem cell or solid organ transplantation.
27. History of severe allergic anaphylactic reactions to chimeric human or humanized antibodies, or fusion proteins.
28. Known hypersensitivity to CHO cell products or any component of the atezolizumab formulation.
29. Uncontrolled intercurrent illness including, but not limited to, psychiatric illness/social situations that in the opinion of the Investigator would compromise compliance to study requirements or put the patient at unacceptable risk.
30. Other malignancy within the past 2 years (not including basal cell or squamous cell carcinoma of the skin, prostate cancer without the need of other treatment than hormones or in situ cervix, breast or melanoma).
31. Live, attenuated vaccines (e.g., FluMist®) are prohibited within 4 weeks prior to initiation of study treatment, during treatment, and for 5 months after the final dose of atezolizumab and/or LOAd703.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angelica Loskog, PhD, Study Chair — Lokon Pharma AB
Locations (3):
- United States (2):
  - Cedars-Sinai Medical Center, The Angeles Clinic and Research Institute, Los Angeles, California
  - Baylor St Luke's Medical Center, Houston, Texas
- Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Overall, a total of 26 subjects signed the informed consent, 2 out of 26 subjects were screening failures and 24 out of 26 subjects were enrolled in the study.
Groups:
- Group 1 LOAd703 1x10e11 VP Plus Atezolizumab: Delolimogene mupadenorepvec (1x10e11 VP) plus atezolizumab
  delolimogene mupadenorepvec: LOAd703 is an oncolytic adenovirus encoding TMZ-CD40L and 4-1BBL
  atezolizumab: Atezolizumab is an anti-PD-L1 antibody
- Group 2 LOAd703 5x10e11 VP Plus Atezolizumab: Delolimogene mupadenorepvec (5x10e11 VP) plus atezolizumab
  delolimogene mupadenorepvec: LOAd703 is an oncolytic adenovirus encoding TMZ-CD40L and 4-1BBL
  atezolizumab: Atezolizumab is an anti-PD-L1 antibody
Period: Group 1: LOAd703 Dose Level 1x10e11 VP
Arm/Group | Group 1 LOAd703 1x10e11 VP Plus Atezolizumab | Group 2 LOAd703 5x10e11 VP Plus Atezolizumab
Started | 7 | 0
Completed | 3 | 0
Not Completed | 4 | 0
Not completed — Death | 4 | 0
Period: Group 2: LOAd703 Dose Level 5x10e11 VP
Arm/Group | Group 1 LOAd703 1x10e11 VP Plus Atezolizumab | Group 2 LOAd703 5x10e11 VP Plus Atezolizumab
Started | 0 | 17
Completed | 0 | 8
Not Completed | 0 | 9
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Death | 0 | 7
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 LOAd703 1x10e11 VP Plus Atezolizumab | Group 2 LOAd703 5x10e11 VP Plus Atezolizumab | Total
Number analyzed (Participants) | 7 | 17 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (10.2) | 60.0 (13.4) | 61.5 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 9 | 11
  Male | 5 | 8 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 7 | 12 | 19
  Unknown or Not Reported | 0 | 4 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 7 | 14 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  Sweden | 5 | 12 | 17
  United States | 2 | 5 | 7
Disease stage at initial diagnosis [Count of Participants; unit: Participants] — Stage 0 melanoma in situ; Stage I Melanoma (localized tumor, up to 2mm by Breslow depth); Stage II Melanoma (localized tumor); Stage III Melanoma (regional spread); Stage IV Melanoma (metastasis beyond regional lymph nodes). Stages I and II: overall favorable prognosis; Stage III: prognosis rather heterogeneous; Stage IV: poor prognosis
  Participants
    Stage 0 | 0 | 1 | 1
    Stage I | 2 | 3 | 5
    Stage II | 0 | 2 | 2
    Stage III | 4 | 8 | 12
    Stage IV | 1 | 2 | 3
    Unknown | 0 | 1 | 1
Disease stage at study entry [Count of Participants; unit: Participants] — Stage 0 melanoma in situ; Stage I Melanoma (localized tumor, up to 2mm by Breslow depth); Stage II Melanoma (localized tumor); Stage III Melanoma (regional spread); Stage IV Melanoma (metastasis beyond regional lymph nodes).
  Stages I and II: overall favorable prognosis; Stage III: prognosis rather heterogeneous; Stage IV: poor prognosis
  Participants
    Stage III | 0 | 0 | 0
    Stage IV | 7 | 17 | 24
    Unknown | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Tolerability Evaluated by NCI CTCAE v5.0
Description: The AE reporting period begins upon receiving the first LOAd703 and/or atezolizumab treatment and continues until final visit at week 57
Time Frame: Up to 57 weeks post treatment initiation
Measure: Number; unit: Number of Events
Arm/Group | Group 1 LOAd703 1x10e11 VP Plus Atezolizumab | Group 2 LOAd703 5x10e11 VP Plus Atezolizumab
Number analyzed (Participants) | 7 | 17
Number of Events
  All Adverse Events (AEs) | 52 | 130
  All Serious Adverse Events (SAEs) | 6 | 11
  Serious Adverse Reactions (SARs) Related to LOAd703 | 0 | 2
  Serious Adverse Reactions (SARs) Related to Atezolizumab | 0 | 1
  AEs Leading to Withdrawal from the Study | 0 | 0
  AEs Leading to LOAd703 Discontinuation | 4 | 4
  AEs Leading to Atezolizumab Discontinuation | 6 | 4
  AEs Leading to Death | 1 | 0
  AEs Related to LOAd703 | 28 | 64
  AEs Related to Atezolizumab | 20 | 41
  AEs Related to LOAd703 and/or Atezolizumab | 30 | 72
  AEs Related to LOAd703 - Grade 1 | 17 | 40
  AEs Related to LOAd703 - Grade 2 | 11 | 22
  AEs Related to LOAd703 - Grade 3 | 0 | 2
  AEs Related to LOAd703 - Grade 4 | 0 | 0
  AEs Related to LOAd703 - Grade 5 | 0 | 0
  AEs Related to Atezolizumab - Grade 1 | 10 | 26
  AEs Related to Atezolizumab - Grade 2 | 10 | 14
  AEs Related to Atezolizumab - Grade 3 | 0 | 1
  AEs Related to Atezolizumab - Grade 4 | 0 | 0
  AEs Related to Atezolizumab - Grade 5 | 0 | 0
  AEs Not Related to LOAd703 or Atezolizumab - Grade 1 | 7 | 32
  AEs Not Related to LOAd703 or Atezolizumab - Grade 2 | 7 | 13
  AEs Not Related to LOAd703 or Atezolizumab - Grade 3 | 7 | 11
  AEs Not Related to LOAd703 or Atezolizumab - Grade 4 | 0 | 2
  AEs Not Related to LOAd703 or Atezolizumab - Grade 5 | 1 | 0

2. Secondary Outcome: Overall Response Rate
Description: Tumor size evaluations accordingly to RECIST 1.1.Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable disease (SD), Neither PR nor progressive disease, Progressive disease (PD), >20% increase in the sum of the longest diameter of target lesions. Overall Response (OR) = number of participants with CR or PR.
Time Frame: Up to 57 weeks post treatment initiation
Population: ORR was evaluated in participants receiving at least 3 doses of LOAd703 and/or atezolizumab with available tumor assessment data.
  Group 1 (1x10e11 VP): from a total of 7 participants, 6 met the criteria to be included in this analysis Group 2 (5x10e11 VP): from a total of 17 participants, 15 met the criteria to be included in this analysis
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Group 1 LOAd703 1x10e11 VP Plus Atezolizumab | Group 2 LOAd703 5x10e11 VP Plus Atezolizumab
Number analyzed (Participants) | 6 | 15
Percentage of Participants | 16.7 [0.4 to 64.1] | 20.0 [4.3 to 48.1]

3. Secondary Outcome: Overall Survival
Description: Survival status of patients. Overall survival is defined as the time from the first dose of study treatment (LOAd703 and/or atezolizumab) until death.
Time Frame: From treatment initiation until last patient last visit, assessed up till 36 months
Population: OS was evaluated in participants receiving at least 3 doses of LOAd703 and/or atezolizumab with available tumor assessment data.
  Group 1 (1x10e11 VP): from a total of 7 participants, 6 met the criteria to be included in this analysis Group 2 (5x10e11 VP): from a total of 17 participants, 15 met the criteria to be included in this analysis
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Group 1 LOAd703 1x10e11 VP Plus Atezolizumab | Group 2 LOAd703 5x10e11 VP Plus Atezolizumab
Number analyzed (Participants) | 6 | 15
Months | 26.05 [2.10 to NA] — The maximum CI was not estimated (insufficient number of participants with events). | NA [3.55 to NA] — Median OS, maximum CI was not reached (insufficient number of participants with events).

4. Secondary Outcome: Antibodies Against LOAd703
Description: Fold change between baseline and evaluation visit for anti-adenovirus antibodies (LOAd703).
  The baseline is the last available measurement taken before the first LOAd703 treatment. Evaluation is a measurement taken from subjects receiving at least 3 LOAd703 treatments.
Time Frame: Up to 57 weeks post treatment initiation
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | Group 1 LOAd703 1x10e11 VP Plus Atezolizumab | Group 2 LOAd703 5x10e11 VP Plus Atezolizumab
Number analyzed (Participants) | 5 | 12
fold change | 9.05 (1.73) | 15.86 (9.81)

5. Secondary Outcome: Immune Cell Phenotype
Description: The ratio for CD8+/Treg cells analyzed in blood at baseline and evaluation visit as determined by flow cytometry.
  The baseline is the last available measurement taken before the first LOAd703 treatment. Evaluation is a measurement taken from subjects receiving at least 3 LOAd703 treatments.
Time Frame: Up to 57 weeks post treatment initiation
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Group 1 LOAd703 1x10e11 VP Plus Atezolizumab - Baseline; Group 1 LOAd703 1x10e11 VP Plus Atezolizumab - Evaluation: Delolimogene mupadenorepvec (1x10e11 VP) plus atezolizumab
  delolimogene mupadenorepvec: LOAd703 is an oncolytic adenovirus encoding TMZ-CD40L and 4-1BBL
  atezolizumab: Atezolizumab is an anti-PD-L1 antibody
- Group 2 LOAd703 5x10e11 VP Plus Atezolizumab - Baseline; Group 2 LOAd703 5x10e11 VP Plus Atezolizumab - Evaluation: Delolimogene mupadenorepvec (5x10e11 VP) plus atezolizumab
  delolimogene mupadenorepvec: LOAd703 is an oncolytic adenovirus encoding TMZ-CD40L and 4-1BBL
  atezolizumab: Atezolizumab is an anti-PD-L1 antibody
Arm/Group | Group 1 LOAd703 1x10e11 VP Plus Atezolizumab - Baseline | Group 2 LOAd703 5x10e11 VP Plus Atezolizumab - Baseline | Group 1 LOAd703 1x10e11 VP Plus Atezolizumab - Evaluation | Group 2 LOAd703 5x10e11 VP Plus Atezolizumab - Evaluation
Number analyzed (Participants) | 4 | 11 | 4 | 11
ratio | 7.63 (1.42) | 14.86 (10.36) | 8.11 (1.23) | 25.37 (20.15)

6. Secondary Outcome: Virus Shedding
Description: Number of samples analyzed that were positive for virus particles in shedding samples.
Time Frame: Up to 57 weeks post treatment initiation
Measure: Number; unit: number of samples
Groups:
- Group 1 LOAd703 1x10e11 VP Plus Atezolizumab - Urine Sample: Delolimogene mupadenorepvec (1x10e11 VP) plus atezolizumab
  delolimogene mupadenorepvec: LOAd703 is an oncolytic adenovirus encoding TMZ-CD40L and 4-1BBL
  atezolizumab: Atezolizumab is an anti-PD-L1 antibody
  Urine shedding
- Group 2 LOAd703 5x10e11 VP Plus Atezolizumab - Urine Sample: Delolimogene mupadenorepvec (5x10e11 VP) plus atezolizumab
  delolimogene mupadenorepvec: LOAd703 is an oncolytic adenovirus encoding TMZ-CD40L and 4-1BBL
  atezolizumab: Atezolizumab is an anti-PD-L1 antibody
  Urine shedding
- Group 1 LOAd703 1x10e11 VP Plus Atezolizumab - Oral Sample: Delolimogene mupadenorepvec (1x10e11 VP) plus atezolizumab
  delolimogene mupadenorepvec: LOAd703 is an oncolytic adenovirus encoding TMZ-CD40L and 4-1BBL
  atezolizumab: Atezolizumab is an anti-PD-L1 antibody
  Oral shedding
- Group 2 LOAd703 5x10e11 VP Plus Atezolizumab - Oral Sample: Delolimogene mupadenorepvec (5x10e11 VP) plus atezolizumab
  delolimogene mupadenorepvec: LOAd703 is an oncolytic adenovirus encoding TMZ-CD40L and 4-1BBL
  atezolizumab: Atezolizumab is an anti-PD-L1 antibody
  Oral shedding
- Group 1 LOAd703 1x10e11 VP Plus Atezolizumab - Rectal Sample: Delolimogene mupadenorepvec (1x10e11 VP) plus atezolizumab
  delolimogene mupadenorepvec: LOAd703 is an oncolytic adenovirus encoding TMZ-CD40L and 4-1BBL
  atezolizumab: Atezolizumab is an anti-PD-L1 antibody
  Rectal shedding
- Group 2 LOAd703 5x10e11 VP Plus Atezolizumab - Rectal Sample: Delolimogene mupadenorepvec (5x10e11 VP) plus atezolizumab
  delolimogene mupadenorepvec: LOAd703 is an oncolytic adenovirus encoding TMZ-CD40L and 4-1BBL
  atezolizumab: Atezolizumab is an anti-PD-L1 antibody
  Rectal shedding
Arm/Group | Group 1 LOAd703 1x10e11 VP Plus Atezolizumab - Urine Sample | Group 2 LOAd703 5x10e11 VP Plus Atezolizumab - Urine Sample | Group 1 LOAd703 1x10e11 VP Plus Atezolizumab - Oral Sample | Group 2 LOAd703 5x10e11 VP Plus Atezolizumab - Oral Sample | Group 1 LOAd703 1x10e11 VP Plus Atezolizumab - Rectal Sample | Group 2 LOAd703 5x10e11 VP Plus Atezolizumab - Rectal Sample
Number analyzed (Participants) | 7 | 17 | 7 | 17 | 7 | 17
number of samples | 0 | 2 | 0 | 1 | 0 | 1

7. Secondary Outcome: Overall Survival (Number of Participants With Event)
Description: Survival status of patients described by number of participants with event.
Time Frame: From treatment initiation until last patient last visit, assessed up till 36 months
Measure: Number; unit: Number of Participants
Arm/Group | Group 1 LOAd703 1x10e11 VP Plus Atezolizumab | Group 2 LOAd703 5x10e11 VP Plus Atezolizumab
Number analyzed (Participants) | 7 | 17
Number of Participants
  Number of Subjects with Event (death) | 4 | 7
  Number of Subjects Censored (at the last date known to be alive) | 3 | 10

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the first LOAd703 and/or atezolizumab treatment up to final clinical follow-up visit at Week 57. All-Cause Mortality was assessed from treatment initiation until last patient last visit, up till 36 months.
Description: The number of participants with adverse events and not the number of events are reported.
Arm/Group | Group 1 LOAd703 1x10e11 VP Plus Atezolizumab | Group 2 LOAd703 5x10e11 VP Plus Atezolizumab
All-Cause Mortality (participants affected / at risk) | 4/7 | 7/17
Serious Adverse Events (participants affected / at risk) | 2/7 | 5/17
Other Adverse Events (participants affected / at risk) | 7/7 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 LOAd703 1x10e11 VP Plus Atezolizumab (N=7) | Group 2 LOAd703 5x10e11 VP Plus Atezolizumab (N=17)
General physical health deterioration (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 1
Salmonellosis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Lymphoedema (Vascular disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cytokine release syndrome (Immune system disorders) | 0 | 1
Medication error (Injury, poisoning and procedural complications) | 0 | 1
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 LOAd703 1x10e11 VP Plus Atezolizumab (N=7) | Group 2 LOAd703 5x10e11 VP Plus Atezolizumab (N=17)
Pyrexia (General disorders) | 4 | 11
Fatigue (General disorders) | 1 | 5
Chills (General disorders) | 2 | 3
Injection site pain (General disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 3 | 5
Vomiting (Gastrointestinal disorders) | 2 | 5
Diarrhoea (Gastrointestinal disorders) | 0 | 4
Nasopharyngitis (Infections and infestations) | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 5
Lymphocyte count decreased (Investigations) | 0 | 2
Headache (Nervous system disorders) | 1 | 4
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 3
Cytokine release syndrome (Immune system disorders) | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 1
Oedema peripheral (General disorders) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Hypotension (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Inflammation (General disorders) | 0 | 1
Injection site reaction (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1
Blood albumin decreased (Investigations) | 0 | 1
Borrelia test positive (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Troponin I increased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Embolism (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-06-09): https://cdn.clinicaltrials.gov/large-docs/70/NCT04123470/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-11): https://cdn.clinicaltrials.gov/large-docs/70/NCT04123470/SAP_001.pdf